CLINICAL TRIAL: NCT04130724
Title: Characterization of a Portable Solid-State Breath Acetone Testing Device for Real-Time Ketosis Status and Comparison to Blood Ketone Testing
Brief Title: Characterization of a Portable Solid-State Breath Acetone Testing Device for Real-Time Ketosis Status
Status: Completed | Type: Observational
Sponsor: Readout, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-0001
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Ketogenic Dieting; Ketosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Ketogenic diet: Subjects consuming either a ketogenic (<30g carbohydrate per day) or a low-carb (<100g carbohydrate per day) diet.
  Interventions: Diagnostic Test: Blood ketone testing; Diagnostic Test: Breath ketone testing
- High-carbohydrate diet: Subjects consuming a high carbohydrate (>100g carbohydrate per day) diet.
  Interventions: Diagnostic Test: Blood ketone testing; Diagnostic Test: Breath ketone testing

INTERVENTIONS:
Diagnostic Test: Blood ketone testing — Ketone testing will be done using a blood beta-hydroxybutyrate (BHB) test at least five (5) times per day.
  Other Names: Blood ketone testing using the Abbott Precision Xtra meter.
Diagnostic Test: Breath ketone testing — Ketone testing will be done using a breath acetone (BrAce) test at least five (5) times per day.
  Other Names: Breath ketone testing using the Readout breath acetone device.

SUMMARY:
The primary purpose of this study is to characterize the performance and utility of a novel breath acetone meter developed by Readout, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Ketogenic diet cohort: currently following a ketogenic or low-carbohydrate diet defined as less than 30 grams per day (ketogenic) or less than 100 grams per day (low-carbohydrate) as estimated by the individual. Subjects must have been following the diet before the beginning of the study period and must continue with the diet throughout the duration of the trial.
* High-carbohydrate diet cohort: currently following a diet that does not restrict dietary carbohydrate. Carbohydrate consumption should be greater than 100 grams per day as estimated by the individual. Subjects must have been following the diet before the study period and must continue with the diet throughout the duration of the trial.

Exclusion Criteria:

* Type-1 diabetes
* Insulin-dependent type-2 diabetes
* History of diabetic ketoacidosis
* Currently taking Warfarin or other blood thinners
* Currently taking a sodium-glucose cotransporter-2 (SGLT2) inhibitor
* Currently taking Disulfiram
* Unwilling to maintain their diet during the study period
* Unwilling to test blood and breath ketones five times per day
* Non-English speaking
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are interested in the ketogenic diet or in tracking their ketones.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Correlation between breath acetone (BrAce) and blood beta-hydroxybutyrate (BHB) concentrations | 2 weeks
  Blood BHB and BrAce measurements will be taken simultaneously during at least five (5) measurement sessions each day. After aggregating data from all study participants, the correlation between these two measurements will be determined using regression analysis.

SECONDARY OUTCOMES:
Reliability of the Readout breath acetone device | 2 weeks
  Multiple BrAce measurements will be taken during each measurement session using the Readout BrAce device and repeatability will be analyzed using alpha reliability coefficients.

OTHER OUTCOMES:
Utility of a single ketone measurement compared to multiple measurements throughout the day | 2 weeks
  The utility of a single BrAce measurement compared to multiple measurements throughout the day will be assessed by comparing a single measurement for a given user with the time-weighted average of all measurements taken that same day. The probability that a single measurement differs from the time-weighted average of all measurements during the same day will be computed for various difference thresholds.
Time dynamics of breath acetone compared to blood beta-hydroxybutyrate | 2 weeks
  The time dynamics of blood BHB versus BrAce will be explored by performing a correlation calculation between the two measurement methods for various time shifts.
Full-day ketone exposure as measured by breath acetone and blood beta-hydroxybutyrate | 2 weeks
  The full-day ketone exposure as measured by BrAce will be compared with the full-day ketone exposure as measured by blood BHB (12 AM on day 1 to 12 AM on day 2) by first performing linear interpolation between data points on a given day and then calculating the daily area under the curve (AUC) for BrAce and blood BHB. The correlation between blood and breath AUC will be determined by performing regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: James McCarter, MD, PhD, Principal Investigator — Readout, Inc.
Locations (1):
- Center for Emerging Technologies, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hallberg SJ, McKenzie AL, Williams PT, Bhanpuri NH, Peters AL, Campbell WW, Hazbun TL, Volk BM, McCarter JP, Phinney SD, Volek JS. Effectiveness and Safety of a Novel Care Model for the Management of Type 2 Diabetes at 1 Year: An Open-Label, Non-Randomized, Controlled Study. Diabetes Ther. 2018 Apr;9(2):583-612. doi: 10.1007/s13300-018-0373-9. Epub 2018 Feb 7. PMID 29417495
- [Background] Bhanpuri NH, Hallberg SJ, Williams PT, McKenzie AL, Ballard KD, Campbell WW, McCarter JP, Phinney SD, Volek JS. Cardiovascular disease risk factor responses to a type 2 diabetes care model including nutritional ketosis induced by sustained carbohydrate restriction at 1 year: an open label, non-randomized, controlled study. Cardiovasc Diabetol. 2018 May 1;17(1):56. doi: 10.1186/s12933-018-0698-8. PMID 29712560
- [Background] Evert AB, Dennison M, Gardner CD, Garvey WT, Lau KHK, MacLeod J, Mitri J, Pereira RF, Rawlings K, Robinson S, Saslow L, Uelmen S, Urbanski PB, Yancy WS Jr. Nutrition Therapy for Adults With Diabetes or Prediabetes: A Consensus Report. Diabetes Care. 2019 May;42(5):731-754. doi: 10.2337/dci19-0014. Epub 2019 Apr 18. No abstract available. PMID 31000505
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Van Gaal L, Scheen A. Weight management in type 2 diabetes: current and emerging approaches to treatment. Diabetes Care. 2015 Jun;38(6):1161-72. doi: 10.2337/dc14-1630. PMID 25998297
- [Background] Boden G, Sargrad K, Homko C, Mozzoli M, Stein TP. Effect of a low-carbohydrate diet on appetite, blood glucose levels, and insulin resistance in obese patients with type 2 diabetes. Ann Intern Med. 2005 Mar 15;142(6):403-11. doi: 10.7326/0003-4819-142-6-200503150-00006. PMID 15767618
- [Background] Shimazu T, Hirschey MD, Newman J, He W, Shirakawa K, Le Moan N, Grueter CA, Lim H, Saunders LR, Stevens RD, Newgard CB, Farese RV Jr, de Cabo R, Ulrich S, Akassoglou K, Verdin E. Suppression of oxidative stress by beta-hydroxybutyrate, an endogenous histone deacetylase inhibitor. Science. 2013 Jan 11;339(6116):211-4. doi: 10.1126/science.1227166. Epub 2012 Dec 6. PMID 23223453
- [Background] Anderson JC. Measuring breath acetone for monitoring fat loss: Review. Obesity (Silver Spring). 2015 Dec;23(12):2327-34. doi: 10.1002/oby.21242. Epub 2015 Nov 2. PMID 26524104
- [Background] Musa-Veloso K, Likhodii SS, Cunnane SC. Breath acetone is a reliable indicator of ketosis in adults consuming ketogenic meals. Am J Clin Nutr. 2002 Jul;76(1):65-70. doi: 10.1093/ajcn/76.1.65. PMID 12081817